CLINICAL TRIAL: NCT02642965
Title: A Phase 1/2 Study of CPX-351 (NSC# 775341) Alone Followed by Fludarabine, Cytarabine, and G-CSF (FLAG) for Children With Relapsed Acute Myeloid Leukemia (AML)
Brief Title: Liposome-encapsulated Daunorubicin-Cytarabine, Fludarabine Phosphate, Cytarabine, and Filgrastim in Treating Younger Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAML1421; NCI-2015-01917 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML1421; PAAML1421_R02PAPP01; s16-00955; AAML1421 (Other: Children's Oncology Group); AAML1421 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2015-12-02; First posted 2015-12-30 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia Post Cytotoxic Therapy; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: interventions — Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine phosphate; CPX-351; Injections; Daunorubicin; Liposomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (CPX-351 and FLAG) (Experimental): COURSE 1: Patients receive cytarabine IT on day 0 and at day 28-30 or up to 7 days prior to day 1 of course 2, and liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5. Patients with CNS1 receive no further CNS-directed therapy in course 1. Patients with CNS2 disease may receive additional 4-6 doses of cytarabine IT twice weekly starting 48 hours after the third dose of liposome-encapsulated daunorubicin-cytarabine until CNS is clear at the discretion of the investigator. Patients meeting criteria for CR, CRp, and CRi may proceed to course 2.
  COURSE 2: Patients receive filgrastim on days 1-5 and then on day 15 until blood count recovery, and fludarabine phosphate IV over 30 minutes and high-dose cytarabine IV over 1-3 hours QD on days 1-5.
  Interventions: Drug: Cytarabine; Biological: Filgrastim; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Filgrastim — Given SC or IV
  Other Names: Filgrastim-aafi; Filgrastim-ayow; G-CSF; Neupogen; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tevagrastim
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of liposome-encapsulated daunorubicin-cytarabine when given with fludarabine phosphate, cytarabine, and filgrastim and to see how well they work in treating younger patients with acute myeloid leukemia that has come back after treatment (relapsed) or is not responding to treatment (is refractory). Liposome-encapsulated daunorubicin-cytarabine is made up of two chemotherapy drugs, cytarabine and daunorubicin hydrochloride, and works to stop cancer cell growth by blocking the cells from dividing. Drugs used in chemotherapy, such as fludarabine phosphate and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Filgrastim may increase the production of blood cells and may help the immune system recover from the side effects of chemotherapy. Giving liposome-encapsulated daunorubicin-cytarabine followed by fludarabine phosphate, cytarabine, and filgrastim may be a better treatment for patients with relapsed acute myeloid leukemia and may cause fewer side effects to the heart, a common effect of other chemotherapy treatments for acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine a recommended phase 2 dose (RP2D) and the toxicities associated with liposome-encapsulated daunorubicin-cytarabine (CPX-351) in pediatric and young adult patients with relapsed/refractory acute myeloid leukemia (AML).

II. To estimate the response rate (complete remission [CR] plus complete remission with partial platelet recovery [CRp]) after CPX-351 (cycle 1) followed by fludarabine phosphate, cytarabine, and filgrastim (FLAG) (cycle 2) in children with AML in first relapse.

SECONDARY OBJECTIVES:

I. To estimate the response rate (CR + CRp + complete remission with incomplete blood count recovery [CRi]) after one cycle of CPX-351.

II. To describe the pharmacokinetics of plasma cytarabine and daunorubicin after CPX-351 administration to pediatric and young adult patients with relapsed/refractory AML.

TERTIARY OBJECTIVES:

I. To describe the response in biomarkers of cardiac injury to a single cycle of CPX-351.

II. To explore the effect of CPX-351 on novel biochemical and imaging markers of cardiotoxicity, including plasma micro ribonucleic acid (RNAs) (miRNA) and myocardial deformation.

III. To explore the role of rare coding variants as risk factors for anthracycline-induced cardiomyopathy.

OUTLINE:

COURSE 1: Patients receive cytarabine intrathecally (IT) on day 0 and at day 28-30 or up to 7 days prior to day 1 of course 2, and liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5. Patients without evidence of central nervous system (CNS) disease (CNS1) receive no further CNS-directed therapy in course 1. Patients with < 5 white blood cells per microliter of blood with blast cells (CNS2) disease may receive additional 4-6 doses of cytarabine IT twice weekly starting 48 hours after the third dose of liposome-encapsulated daunorubicin-cytarabine until CNS is clear at the discretion of the investigator. Patients meeting criteria for CR, CRp, and CRi may proceed to course 2.

COURSE 2: Patients receive filgrastim on days 1-5 and then on day 15 until blood count recovery, and fludarabine phosphate IV over 30 minutes and high-dose cytarabine IV over 1-3 hours once daily (QD) on days 1-5.

After completion of study treatment, patients are followed up periodically for 12 months, and then yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of AML at original diagnosis
* Patient must have one of the following:

  * Recurrent disease with >= 5% blasts in the bone marrow (M2/M3 bone marrow), with or without extramedullary disease.
  * Recurrent disease with an absolute blast count greater than 1,000 per microliter in the peripheral blood with or without extramedullary disease
* To be eligible for the dose-finding phase: (the dose-finding phase completed in 12/2016)

  * Relapsed patients

    * Patients must be in first relapse, and
    * Patients must not have received prior re-induction therapy
  * Refractory patients

    * Patients must not have received more than one attempt at remission induction, which may consist of up to two different therapy courses; Children Oncology Group (COG) AAML1031 de novo therapy including induction I and induction II is an example
  * Treatment-related AML (t-AML)

    * Patients must be previously untreated for secondary AML
* To be eligible for the phase 2 efficacy phase:

  * Relapse patients:

    * Patients must be in first marrow relapse, and
    * Patients must not have received prior re-induction therapy; donor lymphocyte infusion (DLI) is considered a re-induction attempt
* Patients must have the status of CNS1 or CNS2 only, and no clinical signs or neurologic symptoms suggestive of CNS leukemia, such as cranial palsy
* Patients must have a performance status corresponding to an Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age; Note: patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, stem cell transplant or radiotherapy prior to entering this study; all prior treatment-related toxicities must have resolved to =< grade 2 prior to enrollment
* Myelosuppressive chemotherapy: must not have received myelosuppressive chemotherapy within 3 weeks of entry onto this study (excluding hydroxyurea)

  * Cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of CPX-351
* Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biologic agent such as steroids, retinoids; Note: for agents that have known adverse events occurring beyond 7 days after administration (i.e. monoclonal antibodies), this period must be extended beyond the time during which acute adverse events are known to occur
* Radiation therapy (RT): >= 2 weeks for local palliative RT (small port); >= 6 months must have elapsed if prior craniospinal RT or if >= 50% radiation of pelvis; >= 6 weeks must have elapsed if other substantial bone marrow (BM) radiation; Note: patients must have received =< than 13.6 Gray (Gy) prior radiation to the mediastinum
* Stem cell transplant (SCT): no evidence of active graft vs. host disease for at least 4 weeks; for allogeneic SCT patients, >= 3 months must have elapsed since transplant

  * Must have received no more than 1 prior autologous or allogeneic stem cell transplant.
  * Patients must be off all systemic immunosuppressive therapy for at least 2 weeks, excluding hydrocortisone for physiologic cortisol replacement
* Intrathecal cytotoxic therapy:

  * No waiting period is required for patients having received intrathecal cytarabine, methotrexate, and/or hydrocortisone
  * At least 14 days must have elapsed since receiving liposomal cytarabine (DepoCyte) by intrathecal injection
* Growth factors:

  * Patients must not have received growth factors for 7 days prior to CPX-351
  * Patients must not have received pegfilgrastim for 14 days prior to CPX-351
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age 1 to < 2 years: maximum serum creatinine 0.6 mg/dL (males and females)
  * Age 2 to < 6 years: maximum serum creatinine 0.8 mg/dL (males and females)
  * Age 6 to < 10 years: maximum serum creatinine 1.0 mg/dL (males and females)
  * Age 10 to < 13 years: maximum serum creatinine 1.2 mg/dL (males and females)
  * Age 13 to < 16 years: maximum serum creatinine 1.5 mg/dL (males) and 1.4 mg/dL (females)
  * Age >= 16 years: maximum serum creatinine 1.7 mg/dL (males) and 1.4 mg/dL (females)
* Direct bilirubin < 1.5 x upper limit of normal (ULN) for age and institution
* Serum glutamate pyruvate (SGPT) (alanine aminotransferase [ALT]) =< 3.0 x upper limit of normal (ULN) for age and institution (unless it is related to leukemic involvement)
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by radionuclide angiogram or echocardiogram
* Corrected QT (using Bazett's formula [QTcB]) interval < 500 msecs
* Patients with seizure disorder may be enrolled if on anticonvulsants and if seizures are well controlled
* Central nervous system (CNS) toxicity =< grade 2
* Patients with a known history of human immunodeficiency virus (HIV) are eligible, if they meet all of the following conditions:

  * No history of HIV complications with the exception of cluster of differentiation (CD)4 count < 200 cells/mm^3
  * No antiretroviral therapy with overlapping toxicity such as myelosuppression
  * HIV viral loads below the limit of detection
  * No history of highly active antiretroviral therapy (HAART)-resistant HIV
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients who have received > 450 mg/m^2 daunorubicin equivalents; patients who relapse after receiving AAML0531/AAML1031 therapy will be eligible for this study, provided they have not received any additional anthracyclines; NOTE: for the purposes of determining eligibility for this protocol, the following cardiotoxicity multipliers will be used to determine daunorubicin equivalents:

  * Doxorubicin (doxorubicin hydrochloride): 1
  * Mitoxantrone: 3
  * Idarubicin: 3
  * Epirubicin: 0.5
* Patients who are currently receiving another investigational drug
* Patients receiving medications for treatment of left ventricular systolic dysfunction
* Patients with any of the following diagnoses:

  * Acute promyelocytic leukemia (APL)
  * Down syndrome
  * Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome
  * Wilson's disease and any other disorder of copper metabolism
  * Juvenile myelomonocytic leukemia (JMML)
* Patients with documented active, uncontrolled infection at the time of study entry
* Patients with known active hepatitis B virus (HBV) and hepatitis C virus (HCV) infections
* Patients with prior allergy to daunorubicin and/or cytarabine
* Female patients who are pregnant are ineligible
* Lactating females are not eligible
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation and for 6 months after the last dose of chemotherapy

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Cooper, Principal Investigator — Children's Oncology Group
Locations (73):
- United States (67):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital, Asheville, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec

REFERENCES:
- [Derived] Cooper TM, Absalon MJ, Alonzo TA, Gerbing RB, Leger KJ, Hirsch BA, Pollard J, Razzouk BI, Aplenc R, Kolb EA. Phase I/II Study of CPX-351 Followed by Fludarabine, Cytarabine, and Granulocyte-Colony Stimulating Factor for Children With Relapsed Acute Myeloid Leukemia: A Report From the Children's Oncology Group. J Clin Oncol. 2020 Jul 1;38(19):2170-2177. doi: 10.1200/JCO.19.03306. Epub 2020 May 13. PMID 32401633
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (CPX-351 and FLAG)
Started | 38
Completed | 25
Not Completed | 13
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 9

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 26
  More than one race | 1
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 36
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-limiting Toxicity
Description: Number of patients in the dose-finding phase with a dose-limiting toxicity, graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: 28 days
Population: First 6 patients evaluable for dose limiting toxicity (DLT).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Percentage of Responders (Complete Response or Complete Remission With Partial Platelet Recovery) After up to 2 Cycles
Description: Best response (complete response or complete remission with partial platelet recovery) after up to 2 cycles of therapy, where response is assessed using the revised Acute Myeloid Leukemia International Working Group Criteria. Percentage of responders is calculated using the methods of Jung and Kim. 90% confidence interval is determined using the methods of Koyama and Chen.
Time Frame: Up to 8 weeks
Population: 1 patient among the 38 eligible patients was not evaluable for response.
Measure: Number (90% Confidence Interval); unit: Percantage of best responders
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 37
Percantage of best responders | 68.30 [52.89 to 78.02]

3. Secondary Outcome: Percentage of Responders (Complete Response or Complete Remission With Partial or Incomplete Platelet Recovery) After First Cycle of Therapy
Description: Response (complete response or complete remission with partial or incomplete platelet recovery) after first cycle of therapy, where response is assessed using the revised Acute Myeloid Leukemia International Working Group Criteria. Percentage of responders is calculated by the total of number of patients with complete response or complete remission with partial or incomplete platelet recovery divided by the number of patients evaluable for response after the first cycle. 95% confidence interval is determined using a binomial exact method.
Time Frame: Up to 4 weeks
Population: 1 patient among the 38 eligible patients was not evaluable for response.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 37
Percentage of responders | 75.68 [58.80 to 88.23]

4. Secondary Outcome: Liposome-encapsulated Daunorubicin Clearance
Description: Geometric mean liposome-encapsulated daunorubicin clearance following IV infusion will be determined for patients in the dose-finding phase.
Time Frame: Prior to infusion on day 5 and, 45 and 90 minutes post day 5 infusion of cycle 1
Population: Patients in the efficacy phase excluded (n=32). 1 dose finding patient excluded because dose record was not consistent with treatment plan.
Measure: Geometric Mean (Full Range); unit: MILLILITER / HOUR
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 5
MILLILITER / HOUR | 94.7 [47.5 to 193.0]

5. Secondary Outcome: Liposome-encapsulated Daunorubicin Volume of Distribution
Description: Geometric mean liposome-encapsulated daunorubicin volume of distribution following IV infusion will be determined for patients in the dose-finding phase.
Time Frame: Prior to infusion on day 5 and, 45 and 90 minutes post day 5 infusion of cycle 1
Population: as for outcome 4
Measure: Geometric Mean (Full Range); unit: MILLILITER
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 5
MILLILITER | 3827.7 [2165.0 to 6596.0]

6. Secondary Outcome: Liposome-encapsulated Daunorubicin Time of Maximum Concentration
Description: Median liposome-encapsulated daunorubicin time of maximum observed plasma concentration will be determined for patients in the dose-finding phase.
Time Frame: Prior to infusion on day 5 and, 45 and 90 minutes post day 5 infusion of cycle 1
Population: as for outcome 4
Measure: Median (Full Range); unit: HOUR
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 5
HOUR | 2 [1.42 to 2.07]

7. Secondary Outcome: Liposome-encapsulated Daunorubicin Area Under the Curve
Description: Geometric mean liposome-encapsulated daunorubicin area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration will be determined for patients in the dose-finding phase.
Time Frame: Prior to infusion on day 5 and, 45 and 90 minutes post day 5 infusion of cycle 1
Population: as for outcome 4
Measure: Geometric Mean (Full Range); unit: (NANOGRAM x HOUR) / MILLILITER
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 5
(NANOGRAM x HOUR) / MILLILITER | 1288010.3 [761251.0 to 1715266.0]

8. Secondary Outcome: Liposome-encapsulated Cytarabine Clearance
Description: Geometric mean liposome-encapsulated cytarabine clearance following IV infusion will be determined for patients in the dose-finding phase.
Time Frame: Prior to infusion on day 5 and, 45 and 90 minutes post day 5 infusion of cycle 1
Population: as for outcome 4
Measure: Geometric Mean (Full Range); unit: MILLILITER / HOUR
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 5
MILLILITER / HOUR | 71.76 [37.5 to 151.0]

9. Secondary Outcome: Liposome-encapsulated Cytarabine Volume of Distribution
Description: Geometric mean liposome-encapsulated cytarabine volume of distribution following IV infusion will be determined for patients in the dose-finding phase.
Time Frame: Prior to infusion on day 5 and, 45 and 90 minutes post day 5 infusion of cycle 1
Population: as for outcome 4
Measure: Geometric Mean (Full Range); unit: MILLILITER
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 5
MILLILITER | 4158.0 [2642.0 to 7081.0]

10. Secondary Outcome: Liposome-encapsulated Cytarabine Time of Maximum Concentration
Description: Median liposome-encapsulated cytarabine time of maximum observed plasma concentration will be determined for patients in the dose-finding phase.
Time Frame: Prior to infusion on day 5 and, 45 and 90 minutes post day 5 infusion of cycle 1
Population: as for outcome 4
Measure: Median (Full Range); unit: HOUR
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 5
HOUR | 5 [1.92 to 5.07]

11. Secondary Outcome: Liposome-encapsulated Cytarabine Area Under the Curve
Description: Geometric mean liposome-encapsulated cytarabine area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration will be determined for patients in the dose-finding phase.
Time Frame: Prior to infusion on day 5 and, 45 and 90 minutes post day 5 infusion of cycle 1
Population: as for outcome 4
Measure: Geometric Mean (Full Range); unit: (NANOGRAM x HOUR) / MILLILITER
Arm/Group | Treatment (CPX-351 and FLAG)
Number analyzed (Participants) | 5
(NANOGRAM x HOUR) / MILLILITER | 4418582.5 [2765108.0 to 6382600.0]

12. Other Pre Specified Outcome: Length of Hospitalization Time
Description: Descriptive statistics will be used to summarize length of hospitalization time.
Time Frame: Up to 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Time to Bone Marrow Count Recovery
Description: Descriptive statistics will be used to summarize bone marrow count recovery.
Time Frame: Up to 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Time to Peripheral Blood Cell Count Recovery
Description: Descriptive statistics will be used to summarize peripheral blood cell count recovery.
Time Frame: Up to 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Proportion of Patients Experiencing Toxicities
Description: Proportion of patients experiencing >= grade 3 non-hematologic toxicities, cardiac toxicities, and infections by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 8 weeks post-treatment
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Troponin Levels
Description: Spearman correlation coefficients will be used to correlate the post-treatment values of troponin with previous cumulative anthracycline dose prior to liposome-encapsulated daunorubicin-cytarabine, change in ejection fraction between pre- and post-liposome-encapsulated daunorubicin-cytarabine baseline assessed by echocardiogram before and after course 1, and change in global longitudinal strain.
Time Frame: Baseline up to day 30
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in N-terminal Pro B-type Natriuretic Peptide (NT-BNP) Levels
Description: Spearman correlation coefficients will be used to correlate the post-treatment values of NT-BNP with previous cumulative anthracycline dose prior to liposome-encapsulated daunorubicin-cytarabine, change in ejection fraction between pre- and post-liposome-encapsulated daunorubicin-cytarabine baseline assessed by echocardiogram before and after course 1, and change in in global longitudinal strain.
Time Frame: Baseline up to day 30
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in High Sensitive C-reactive Protein (HS-CRP) Levels
Description: Spearman correlation coefficients will be used to correlate the post-treatment values of HS-CRP with previous cumulative anthracycline dose prior to liposome-encapsulated daunorubicin-cytarabine, change in ejection fraction between pre- and post-liposome-encapsulated daunorubicin-cytarabine baseline assessed by echocardiogram before and after course 1, and change in in global longitudinal strain.
Time Frame: Baseline up to day 30
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in in Global Longitudinal Strain
Description: A paired t-test will be used to compare the mean global longitudinal strain between the pre-treatment (at relapse) baseline and post-course 1 echocardiogram.
Time Frame: Baseline up to 28 days
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Micro Ribonucleic Acid (miRNA) Using TaqMan miRNA Assays
Description: Plasma miR-29b and -499 fold change from pre-treatment baseline will be determined at each post-treatment time point using the delta-delta-Ct method. The relationship between 6-hour miR-29b and -499 expression and change in left ventricular global longitudinal strain between the pre-cycle and end of cycle 1 echocardiograms will be determined by calculating a Spearman correlation coefficient.
Time Frame: Baseline up to day 30
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: While patients were on Protocol Therapy (up to 8 weeks) or during follow-up (up to 3 years).
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Treatment (CPX-351 and FLAG)
All-Cause Mortality (participants affected / at risk) | 14/38
Serious Adverse Events (participants affected / at risk) | 21/38
Other Adverse Events (participants affected / at risk) | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (CPX-351 and FLAG) (N=38)
Febrile neutropenia (Blood and lymphatic system disorders) | 11
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 5
Fever (General disorders) | 2
Anorectal infection (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 6
Kidney infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Small intestine infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (CPX-351 and FLAG) (N=38)
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Ventricular arrhythmia (Cardiac disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 4
Multi-organ failure (General disorders) | 1
Device related infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 3
Mucosal infection (Infections and infestations) | 2
Periorbital infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 3
Upper respiratory infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Ejection fraction decreased (Investigations) | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 14
GGT increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 1
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 5
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT02642965/Prot_SAP_002.pdf